CLINICAL TRIAL: NCT04807868
Title: AdventHealth Research Institute Non-Alcoholic Fatty Liver Disease Biobank and Registry (AVAIL)
Acronym: AVAIL
Status: Recruiting | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: BPGbio (Industry)
Responsible Party: Sponsor
Other Study IDs: 1628655
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Liver tissue, fasting blood and spot urine will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Biopsy Group: Adults undergoing a standard of care liver biopsy at AdventHealth Central Florida Division for any reason
  Interventions: Procedure: Standard of care liver biopsy; Other: Fibroscan; Other: Biospecimen Collection
- Non-Biopsy Group: Adults without any history of NAFLD
  Interventions: Other: Fibroscan; Other: Biospecimen Collection

INTERVENTIONS:
Procedure: Standard of care liver biopsy — Patients undergoing a standard of care liver biopsy for any reason who are willing to participate will be consented for collecting additional biopsy tissue for research purposes. 1-2 additional biopsy tissue cores will be collected for research. Liver tissue will be biobanked for future use.
  Groups: Biopsy Group
Other: Fibroscan — A FibroScan will be performed to evaluate longitudinal changes in liver fat and fibrosis.
Other: Biospecimen Collection — Blood and urine will be collected.

SUMMARY:
The purpose of this study is to create a resource that will advance research that is focused on discovery of novel therapies, risk stratification, and aggressive interventions for those at highest risk for non-alcoholic fatty liver disease (NAFLD). To achieve this, we will generate a biobank of liver tissue collected during standard of care liver biopsies. Paired blood/urine samples, FibroScan and relevant data will also be collected.

ELIGIBILITY:
Inclusion Criteria

* Females and Males ≥ 18 years of age.
* Understands the procedures and agrees to participate by giving written informed consent.

Biopsy Group Only:

• Scheduled for standard of care liver biopsy for any reason.

Non-Biopsy Group Only:

• BMI ≥ 25, with or without type 2 diabetes, without any level of NAFLD based on: (1) Recent medical history (within 6 months of screening visit). (2) Data collected from participation in a prior research study where they consented to be re-contacted for future studies.

Exclusion Criteria

* Women who are pregnant when referred for a liver biopsy will be excluded.
* Presence of any condition that, in the opinion of the Investigator, compromises participant safety or data integrity or the participant's ability to complete the study.

Otherwise, all eligible patients who consent will be included in AVAIL. If participants in the non-biopsy group are found to have NAFLD based on the FibroScan done for this study, then they will be informed of this and advised to follow up with their physician. Their data will still be part of the registry and analyzed with the biopsy group that is found to have NAFLD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with Non-alcoholic fatty liver disease (NAFLD) and adults without any history of NAFLD.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Creation of a Biobank of Liver Tissue Paired with a Registry of Histological and Clinical Metadata | Baseline

SECONDARY OUTCOMES:
Creation of a Biobank of Blood and Urine Samples Paired with a Registry of Associated Histological and Clinical Metadata | Baseline with annual follow up for up to 5 years
Change in Liver Fat and Fibrosis Over Time ad Measured with FibroScan Controlled Attenuation Parameter and Vibration Controlled Transient Elastography, respectively | Baseline with annual follow up for up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Karen Corbin, PhD, RD, Principal Investigator — Investigator
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States

REFERENCES:
- See also: Website for AdventHealth Translational Research Institute — https://www.adventhealthresearchinstitute.com/research/translational-research